CLINICAL TRIAL: NCT01140217
Title: An Open Label Study to Evaluate the Contraceptive Efficacy and Safety of Norethindrone Acetate Transdermal Delivery System
Brief Title: Efficacy and Safety Study of Norethindrone Acetate Transdermal Delivery System in Contraception
Acronym: Simplify
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NE0906
Record Dates: First submitted 2010-05-18; First posted 2010-06-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Contraceptive Usage
Keywords: contraception; pregnancy
MeSH Terms: conditions — Contraception Behavior | interventions — Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental): Norethindrone Acetate Transdermal Delivery System
  Interventions: Drug: Norethindrone Acetate

INTERVENTIONS:
Drug: Norethindrone Acetate — Norethindrone Acetate Transdermal Delivery System
  Other Names: NEA TDS

SUMMARY:
The purpose of this study is to determine whether NEA TDS is effective in the prevention of pregnancy. The safety of this product will also be evaluated.

DETAILED DESCRIPTION:
An Open Label Study to Evaluate the Contraceptive Efficacy and Safety of Norethindrone Acetate Transdermal Delivery System.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females
* 18-45 years
* Regular, consistent menstrual cycles between 25 and 35 days
* Sexually active and at risk of becoming pregnant

Exclusion Criteria:

* History of infertility
* Known contraindications to progestogen administration
* Pap smear suggestive of a high-grade precancerous lesion(s)
* Clinically significant deviation from normal in any of the screening tests or exams

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1659 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate | 1 year
  The pregnancy rate will be calculated using the Pearl Index that defined as 1300*Number of pregnancies/Number of cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kim E Caramelli, MS, Study Director — Watson Pharmaceuticals, Inc.
Locations (53):
- United States (53):
  - Watson Investigational Site, Birmingham, Alabama
  - Watson Investigational Site, Mobile, Alabama
  - Watson Investigational Site, Montgomery, Alabama
  - Watson Investigational Site, Chandler, Arizona
  - Watson Investigational Site, Little Rock, Arkansas
  - Watson Investigational Site, Garden Grove, California
  - Watson Investigational Site, La Mesa, California
  - Watson Investigational Site, San Diego, California
  - Watson Investigational Site, Denver, Colorado
  - Watson Investigational Site, Newark, Delaware
  - Watson Investigational Site, Washington D.C., District of Columbia
  - Watson Investigational Site, Aventura, Florida
  - Watson Investigational Site, Daytona Beach, Florida
  - Watson Investigational Site, Jacksonville, Florida
  - Watson Investigational Site, Lake Worth, Florida
  - Watson Investigational Site, Miami, Florida
  - Watson Investigational Site, North Miami, Florida
  - Watson Investigational Site, Pinellas Park, Florida
  - Watson Investigational Site, Sarasota, Florida
  - Watson Investigational Site, Atlanta, Georgia
  - Watson Investigational Site, Decatur, Georgia
  - Watson Investigational Site, Sandy Springs, Georgia
  - Watson Investigational Site, Savannah, Georgia
  - Watson Investigational Site, Chicago, Illinois
  - Watson Investigational Site, Overland Park, Kansas
  - Watson Investigational Site, Marrero, Louisiana
  - Watson Investigational Site, New Orleans, Louisiana
  - Watson Investigational Site, Haverhill, Massachusetts
  - Watson Investigational Site, Ann Arbor, Michigan
  - Watson Investigational Site, Kalamazoo, Michigan
  - Watson Investigational Site, Edina, Minnesota
  - Watson Investigational Site, Las Vegas, Nevada
  - Watson Investigational Site, Lawrenceville, New Jersey
  - Watson Investigational Site, Albuquerque, New Mexico
  - Watson Investigational Site, New York, New York
  - Watson Investigational Site, Chapel Hill, North Carolina
  - Watson Investigational Site, New Bern, North Carolina
  - Watson Investigational Site, Raleigh, North Carolina
  - Watson Investigational Site, Cleveland, Ohio
  - Watson Investigational Site, Columbus, Ohio
  - Watson Investigational Site, Medford, Oregon
  - Watson Investigational Site, Philadelphia, Pennsylvania
  - Watson Investigational Site, Columbia, South Carolina
  - Watson Investigational Site, Greer, South Carolina
  - Watson Investigational Site, Hilton Head Island, South Carolina
  - Watson Investigational Site, Nashville, Tennessee
  - Watson Investigational Site, Austin, Texas
  - Watson Investigational Site, Dallas, Texas
  - Watson Investigational Site, Houston, Texas
  - Watson Investigational Site, San Antonio, Texas
  - Watson Investigational Site, Salt Lake City, Utah
  - Watson Investigational Site, Norfolk, Virginia
  - Watson Investigational Site, Seattle, Washington